CLINICAL TRIAL: NCT02603549
Title: Spontaneous Spinal Cerebrospinal Fluid Leaks and Intracranial Hypotension
Brief Title: Pituitary Function and Spontaneous Intracranial Hypotension
Status: Suspended | Type: Observational
Why Stopped: Study protocol needs to be amended. Recruitment is halted until amendment is completed and approved by IRB.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Vivien Bonert, MD, Clinical Director, Pituitary Center, Cedars-Sinai Medical Center
Other Study IDs: Pro39357
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hyperprolactinemia; Spontaneous Intracranial Hypotension
MeSH Terms: conditions — Hyperprolactinemia; Intracranial Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery or Blood Patch
  Interventions: Other: Pituitary panel will be drawn pre-op and post-op for all patients.

INTERVENTIONS:
Other: Pituitary panel will be drawn pre-op and post-op for all patients.

SUMMARY:
Previous research has identified spontaneous cerebral spinal fluid leakage as a cause for spontaneous intracranial hypotension, leading to positional headache patterns. Typical magnetic resonance imaging findings include subdural fluid collections, enhancement of pachymenginges, engorgement of venous structures, pituitary hyperemia, and sagging of the brain (SEEPS). Because pituitary hyperemia has been documented in cases of spontaneous cerebral spinal fluid leakage and is known to mimic a pituitary tumor or hyperplasia, the investigators would like to like to assess the clinical manifestations and neuroimaging abnormalities of SIH patients with regard to the pituitary gland. Specifically, the investigators are looking to analyze the compression of the pituitary stalk and conduct a systemic evaluation of pituitary function in SIH patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age 18 years and older
* Diagnosis of SIH:
* LP
* Brain MRI (SEEPS)

Exclusion Criteria:

* Pregnant and post-partum females
* Nursing mothers
* Patients with potential hyperprolactinemia due to:
* Hypothyroidism,
* Chronic renal disorder
* Liver disease (including cirrhosis)
* Primary or secondary amenorrhea
* Polycystic Ovary Syndrome
* Seizure disorder
* Illicit drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Spontaneous intracranial hypotension (SIH)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the levels of prolactin pre and post treatment | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Bonert, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Schievink WI. Spontaneous spinal cerebrospinal fluid leaks and intracranial hypotension. JAMA. 2006 May 17;295(19):2286-96. doi: 10.1001/jama.295.19.2286. PMID 16705110
- [Background] SCHALTENBRAND G. Normal and pathological physiology of the cerebrospinal fluid circulation. Lancet. 1953 Apr 25;1(6765):805-8. doi: 10.1016/s0140-6736(53)91948-5. No abstract available. PMID 13036182
- [Background] Mokri B. Cerebrospinal fluid volume depletion and its emerging clinical/imaging syndromes. Neurosurg Focus. 2000 Jul 15;9(1):e6. doi: 10.3171/foc.2000.9.1.6. PMID 16859267